CLINICAL TRIAL: NCT04676269
Title: Amnion Bilayer and Stem Cell Combination Therapy on Thin Endometrium Infertile Patients
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, dr. Achmad Kemal Harzif, SpOG (K), Principal Investigator, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 19-10-1202
Record Dates: First submitted 2020-12-02; First posted 2020-12-21 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Cell- and Tissue-Based Therapy
Keywords: Endometrial stem cells; Amnion epithelial stem cells; Amnion bilayer; Thin endometrium; Secondary amenorrhoe

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: None of the participants, gynecologists, statistician, nurses nor of the participant' partners are informed about the treatment groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Amnion only (Sham Comparator): Amnion bilayer as a scaffold to overlay the endometrium, with minor curettage prior to stick the scaffold.
  Interventions: Biological: Amnion only
- Amnion- self endometrium stem cells (EnSC) (Experimental): Amnion bilayer as a scaffold, seeded with endometrium stem cells to regenerate the thin endometrium.
  Interventions: Biological: Amnion - endometrium cells
- Amnion- amnion epithelial stem cells (AESC) (Experimental): Amnion bilayer as a scaffold, seeded with amnion epithelial stem cells to regenerate the thin endometrium.
  Interventions: Biological: Amnion - amnion epithelial cells
- Amnion- co culture self EnSC - AESC (Experimental): Amnion bilayer as a scaffold, seeded with co-culture of endometrium stem cells and amnion epithelial stem cells to regenerate the thin endometrium.
  Interventions: Biological: Amnion-EnSC-AESC

INTERVENTIONS:
Biological: Amnion only — Patients endometrium will be transplanted with amnion only (without seeded cells)
  Arms: Amnion only
Biological: Amnion - endometrium cells — Patients endometrium will be transplanted with amnion seeded with endometrium cells isolated from the patients themselves
  Arms: Amnion- self endometrium stem cells (EnSC)
Biological: Amnion - amnion epithelial cells — Patients endometrium will be transplanted with amnion seeded with amnion epithelial stem cells isolated from other patients' caesarean sectio amnion membrane (tested HLA-DR negative to prevent rejection)
  Arms: Amnion- amnion epithelial stem cells (AESC)
Biological: Amnion-EnSC-AESC — Patients endometrium will be transplanted with amnion seeded with endometrium cells-amnion epithelial stem cells co-culture
  Arms: Amnion- co culture self EnSC - AESC

SUMMARY:
Severe infections or trauma to the endometrial lining causes permanent scars that disrupt the menstrual cycle and lead to conceive failure. Transplantation of biological graft seeded with stem cells is purposed to regenerate and recover the capability of the endometrial lining back into its cycles. Initially, the techniques to isolate and culture the endometrial cells and amnion epithelial stem cells were developed, then the endometrial cells form patients with thin endometrium. Tissue were obtained from hysteroscopic biopsy, weight between 100 µl, while up to 20 µl from the thin endometrium. Tissue were digested using collagenase-1 and cultured using DMEM-F12 added wit epidermal growth factor. Endometrial cells will be characterized to SSUD2, ICAM and BRCP1. Amnion epithelial stem cells (hAESC) will be isolated using collagenase-1 and hyaluronidase. Characterization towards TRA-1-60, SSEA-4, Oct 3/4, and Nanog. In the future, the cells will be co-culture on amnion bilayer, and stained using IHC against α-cadherin, estrogen receptor α, progesterone receptor. Endometrial receptivity (HOXA10, LIF (early secretory) adhesion, VEGF, osteopontin (SPP1) to indicate the pinopodes will be identified using qPCR.The SPP1, target of MIR424 expressed during the receptive phase.

ELIGIBILITY:
Inclusion Criteria:

* Patients with thin endometrium without scar
* Patients with acute thin endometrium post-therapy (medicamentosa)
* Patients who are willing to participate in the study

Exclusion Criteria:

* Patients with thin endometrium due to TB
* Patients with cancer in the reproductive system

Max Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-12-09 (Actual); Primary Completion 2021-07-15 (Estimated); Study Completion 2021-12-15 (Estimated)

PRIMARY OUTCOMES:
Change in endometrium thickness | 7 and 14 days after amnion bilayer seeded with endometrial cells co-cultured with hAESC is transplanted into patient' womb
  Observation by USG
Change in amenorrhea severity | 7 and 14 days after amnion bilayer seeded with endometrial cells co-cultured with hAESC is transplanted into patient' womb
  Patients' report

CONTACTS AND LOCATIONS:
Overall Officials: Achmad Kemal Harzif, MD, Principal Investigator — Faculty of Medicine, Indonesia University
Locations (1):
- RSUPN Cipto Mangunkusumo, Jakarta Pusat, DKI Jakarta, Indonesia